CLINICAL TRIAL: NCT03246269
Title: Normative Values for the German Version of the Montreal Cognitive Assessment (MoCA)
Acronym: MoCA-Norm
Status: Completed | Type: Observational
Sponsor: Andreas Monsch (Other)
Responsible Party: Sponsor-Investigator, Andreas Monsch, PhD, University Hospital, Basel, Switzerland
Organization: University Hospital, Basel, Switzerland (Other)
Other Study IDs: MoCA-Norm
Record Dates: First submitted 2017-08-08; First posted 2017-08-11 (Actual); Last update posted 2018-05-31 (Actual); Status verified 2018-05

CONDITIONS: Cognitive Impairment; Cognitive Decline; Cognition Disorders; Cognitive Symptom; Cognitive Change; Cognitive Deterioration; Cognitive Abnormality; Cognitive Impairment, Mild; Cognition Disorders in Old Age; Dementia; Dementia Alzheimers; Dementia, Alzheimer Type; Dementia, Mild; Dementia of Alzheimer Type
MeSH Terms: conditions — Cognitive Dysfunction; Cognition Disorders; Neurobehavioral Manifestations; Dementia; Alzheimer Disease; Lymphoma, Follicular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MoCA cohort: The German MoCA is administered once to all study participants.
  Interventions: Diagnostic Test: MoCA

INTERVENTIONS:
Diagnostic Test: MoCA

SUMMARY:
This observational cohort study in healthy volunteers establishes normative data for the German version of the Montreal Cognitive Assessment (MoCA) and investigates the possible impacts of demographics on the MoCA total score.

DETAILED DESCRIPTION:
The Montreal Cognitive Assessment (MoCA) is a short tool to evaluate a multitude of cognitive domains (visuospatial / executive functioning, object naming, memory, attention, language, abstraction, orientation). The original English MoCA consistently showed very high sensitivity and specificity in distinguishing patients with mild cognitive impairment from healthy controls. Therefore it is an excellent tool for early recognition of cognitive disorders. Based on a Canadian sample, the MoCA proposes a cut-off-value of 26/30 points. However, there is increasing evidence of intercultural differences in terms of the best cut-off-score. In addition the original version only slightly corrects for possible influences of education - an adjustment for age- or gender-related effects is missing. Therefore, the aim of our study was to investigate the possible impacts of demographics on the MoCA total score and to provide normative values for a German-speaking population.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥65 years
* Education ≥7 years
* Fluency in the German language
* Written informed consent

Exclusion Criteria:

* History of cognitive impairment
* Depression
* Severe sensory or motor impairment interfering with cognitive testing
* Serious somatic disease
* Disease or event affecting the central nervous system
* Cerebrovascular disease
* Regular medication with psychoactive drugs except for benzodiazepines
* Participation in a cognitive study within the last 3 months

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 334 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Montreal Cognitive Assessment (MoCA) - German version | Baseline
  Total score of the MoCA

SECONDARY OUTCOMES:
Mini-Mental State Examination (MMSE) | Baseline
  Total score of the MMSE
Geriatric Depression Scale (GDS) | Baseline
  Total score of the GDS
Consortium to Establish a Registry for Alzheimer's Disease - Neuropsychological Assessment Battery (CERAD-NAB) | Baseline
  Total score of the CERAD-NAB

CONTACTS AND LOCATIONS:
Overall Officials: Alessandra Thomann, MSc, Principal Investigator — Felix Platter Hospital Basel; Nicolai Goettel, MD, Principal Investigator — University Hospital, Basel, Switzerland; Raphael Monsch, MD, Principal Investigator — University Hospital, Basel, Switzerland; Manfred Berres, PhD, Principal Investigator — University of Applied Sciences Koblenz; Andreas Monsch, PhD, Study Chair — Felix Platter Hospital Basel

IPD SHARING:
Plan to Share IPD: Undecided